CLINICAL TRIAL: NCT01505062
Title: A Phase I/IIA Dose Escalation Safety Study of Subretinally Injected SAR421869, Administered to Patients With Retinitis Pigmentosa Associated With Usher Syndrome Type 1B
Brief Title: Study of SAR421869 in Participants With Retinitis Pigmentosa Associated With Usher Syndrome Type 1B
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study stopped not for safety reasons. Due to review of clinical development plans and priorities, Sponsor decided to stop development of the product.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDU13600; US1/001/10 (Other: Oxford Biomedica)
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Usher Syndrome; Retinitis Pigmentosa
Keywords: Usher Syndrome Retinitis Pigmentosa; Usher Syndrome associated Retinitis Pigmentosa
MeSH Terms: conditions — Usher Syndromes; Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- SAR421869 (Cohort 1) (Experimental): Starting dose of SAR421869 given through one subretinal injection.
  Interventions: Drug: SAR421869
- SAR421869 (Cohort 2) (Experimental): Escalating dose of SAR421869 given through one subretinal injection.
  Interventions: Drug: SAR421869
- SAR421869 (Cohort 3) (Experimental): Escalating dose of SAR421869 given through one subretinal injection.
  Interventions: Drug: SAR421869
- SAR421869 (Cohort 4) (Experimental): Maximum tolerated dose (MTD) of SAR421869 given through one subretinal injection.
  Interventions: Drug: SAR421869
- SAR421869 (Cohort 5) (Experimental): MTD of SAR421869 given through one subretinal injection.
  Interventions: Drug: SAR421869

INTERVENTIONS:
Drug: SAR421869 — Formulation: Sterile suspension for intraocular injection, 100 microliters (μL) aliquots in 0.3 milliliter (mL) type I borosilicate glass 'V' vials with a butyl stopper and aluminum crimp seal.
  Route of administration: subretinal injection
  Other Names: UshStat®

SUMMARY:
To evaluate the safety and tolerability of ascending doses of subretinal injections of SAR421869 in participants with Usher syndrome type 1B.

To evaluate for possible biological activity of SAR421869.

DETAILED DESCRIPTION:
Following screening procedures, the gene transfer agent were injected once only under the retina by an opthalmic surgeon under anesthesia. Participants then had regular follow-up visits where general health examinations, blood tests and ophthalmic examinations including best corrected visual acuity, slit lamp examination, intraocular pressure, fundoscopy, autofluorescence, optical coherence tomography, perimetry and electroretinogram were undertaken.

At the end of the study, the participants were invited to enter in an open-label safety study for long-term follow-up visits (at least once every six months) including ophthalmological examinations and recording of adverse events (AEs) were continued for 5 years; then the Investigator followed the participants by telephone for a subsequent 10 years at a minimum interval of once a year to monitor delayed AEs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and molecular diagnosis of Retinitis Pigmentosa associated with Usher Syndrome type 1B, caused by at least one pathogenic myosin 7a gene (MYO7A) mutation on both alleles, confirmed by direct sequencing and co-segregation analysis within the participant's family.
* Suitable verbal/auditory and/or tactile sign language communication (in the opinion of the investigator) as to allow written informed consent to be obtained.
* Women of childbearing potential had a negative pregnancy test at screening and at baseline, and agree to use an effective form of contraception such as the contraceptive pill or intra uterine device for at least three months following SAR421869 administration, or be surgically sterile or postmenopausal, with the last menstrual period being over two years prior to enrolment.
* Males of reproductive potential agreed with their partner to use two forms of contraception, including one barrier method for at least three months following SAR421869 administration if their partner was of childbearing capacity, or must be surgically sterile.
* Participants agreed to not donate blood, organs, tissues or cells for at least three months following SAR421869 administration.

Exclusion Criteria:

* Presence of significant ocular abnormalities in the study eye that in the opinion of the investigator would preclude the planned surgery, effective safety follow-up, or interfere with the interpretation of study outcome measures (e.g., glaucoma, corneal or significant lens opacities, pre-existing uveitis, intraocular infection, choroidal neovascularization).
* Any pre-existing factor or past history of eye disease in children that might predispose to an increased risk of surgical complications in the study eye (e.g., trauma, previous surgery, uveitis, congenital, developmental or structural abnormalities).
* Concomitant systemic diseases including those in which the disease itself, or the treatment for the disease, can alter ocular function (e.g., malignancies, diabetes, juvenile rheumatoid arthritis or sickle cell disease).
* Any contraindication to pupil dilation in either eye.
* Contraindications to use of anesthesia (local or general, as appropriate).
* Treatment with intravitreal, subtenon, or periocular steroid within 4 months of the screening visit.
* Any known allergy to any component of the delivery vehicle or diagnostic agents used during the study (e.g., fluorescein, dilation drops), or medications planned for use during the peri-operative period, particularly topical, injected or systemic corticosteroids.
* Life-threatening illness.
* Alcohol or other substance abuse.
* History of malignancy within a five year period or have had a positive cancer screening test within a one year period of the screening visit.
* Laboratory test abnormalities or abnormalities in electrocardiogram or chest X-ray, that in the opinion of the principal investigator, are clinically significant and would make the participant unsuitable for participation in the study.
* Intercurrent illness or infection 28 days prior to SAR421869 administration.
* Concurrent anti-retroviral therapy that would inactivate the investigational agent.
* Current treatment with immunosuppressant therapies.
* Pre-menopausal or non-surgically sterile women who were unwilling to use an effective form of contraception such as the contraceptive pill or intrauterine device.
* Men or women who did not agree to use barrier contraception as specified in the inclusion criteria.
* Pregnant or breastfeeding women.
* History of any investigational agent within 28 days prior to SAR421869 administration.
* Participation in a prior gene transfer therapy study.
* Enrolment in any other clinical study, for any condition, including those relating to Usher syndrome Type 1B, throughout the duration of the SAR421869 study.
* Current or anticipated treatment with anticoagulant therapy or the use of anticoagulation therapy within the four weeks prior to surgery.
* Past medical history of HIV, or hepatitis A, B or C.
* Inability to comply with the study protocol.
* Any ocular surgery including laser and cataract surgery with intraocular lens implantation, aphakia or prior vitrectomy, in the study eye within 6 months of screening.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Weleber, MD, Principal Investigator — Casey Eye Institute, Portland, Oregon; Jose-Alain Sahel, MD, PhD, Principal Investigator — Hopital Nationale des Quinze-Vingt, Paris France
Locations (2):
- Investigational Site Number 840001, Portland, Oregon, United States
- Investigational Site Number 250001, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Zallocchi M, Binley K, Lad Y, Ellis S, Widdowson P, Iqball S, Scripps V, Kelleher M, Loader J, Miskin J, Peng YW, Wang WM, Cheung L, Delimont D, Mitrophanous KA, Cosgrove D. EIAV-based retinal gene therapy in the shaker1 mouse model for usher syndrome type 1B: development of UshStat. PLoS One. 2014 Apr 4;9(4):e94272. doi: 10.1371/journal.pone.0094272. eCollection 2014. PMID 24705452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In 2017, Sanofi suspended trials of SAR421869, while assessing its future. Until final decision was made, trial TDU13600 was not complete and in fact, further recruitment was planned. In 2019, Sanofi decided to terminate trial due to final decision on SAR421869, and shared decision with health authorities. Results have been reported expeditiously.
Pre-assignment Details: A total of 11 participants were screened. Nine participants of them were enrolled in the study with 3 participants in each of Cohorts 1 to 3. Due to early termination no participant was recruited in Cohorts 4 and 5.
Groups:
- Cohort 1: Participants received subretinally a single injection of SAR421869 at target dose of 1.4*10^5 transducing units (TU) per eye.
- Cohort 2: Participants received subretinally a single injection of SAR421869 at target dose of 4.7*10^5 TU per eye.
- Cohort 3: Participants received subretinally a single injection of SAR421869 at target dose of 1.4*10^6 TU per eye.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population that included all participants who were enrolled in the study and received investigational medicinal product (IMP).
Groups:
- Cohort 1: Participants received subretinally a single injection of SAR421869 at target dose of 1.4*10^5 TU per eye.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Continuous [Median (Full Range); unit: years] | 25 [22 to 28] | 42 [32 to 57] | 50 [32 to 56] | 32 [22 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any unfavorable and unintended physical sign, symptom, or laboratory parameter that developed or worsened in severity during the course of the study, whether or not considered related to the IMP. The TEAEs were defined as any event that started or increased in severity after the participant received IMP, including abnormal laboratory results, electrocardiogram, etc.
Time Frame: From Baseline to Week 48
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
percentage of participants | 100 | 100 | 100

2. Primary Outcome: Percentage of Participants With TEAEs by Severity
Description: An AE was any unfavorable and unintended physical sign, symptom, or laboratory parameter that developed or worsened in severity during the course of the study, whether or not considered related to the IMP. The TEAEs were defined as any event that started or increased in severity after the participant received IMP, including abnormal laboratory results, electrocardiogram, etc. For each AE, the severity was categorized as either mild, moderate or severe where 'mild' was defined as discomfort noticed but did not interfere with the participant's daily routines (an annoyance), 'moderate' was defined as some impairment of function, not hazardous to health (uncomfortable or embarrassing), and 'severe' was defined as significant impairment of function, hazardous to health (incapacitating).
Time Frame: From Baseline to Week 48
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
percentage of participants
  Mild | 100 | 100 | 100
  Moderate | 0 | 33 | 67
  Severe | 0 | 0 | 67

ADVERSE EVENTS:
Time Frame: All AEs were collected from time of first dose of study drug up to Week 48 regardless of seriousness or relationship (causality) to investigational product.
Description: Reported AEs were TEAEs that developed/worsened during the 'on treatment period' (from Day 0 to Week 48). Analysis was performed on safety population.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3)
Uveitis (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3)
Anterior chamber cell (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 3 | 2 | 0
Dyschromatopsia (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 2 | 1 | 1
Eye pruritus (Eye disorders) | 2 | 1 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 1 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1
Subretinal fluid (Eye disorders) | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Injection site extravasation (General disorders) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Intraocular pressure decreased (Investigations) | 1 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 2 | 2
Urine analysis abnormal (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The planned analysis was adjusted and carried out only on the available safety and tolerability data collected before the Sponsor's decision to stop SAR421869 development prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT01505062/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT01505062/SAP_001.pdf